CLINICAL TRIAL: NCT01307748
Title: Physiologic and Expectancy Effects of Stress-reducing Aroma in Older Adults
Brief Title: Effects of Stress-reducing Aromatherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Barry S. Oken, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB#00006890
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Stress-related Problems
Keywords: aromatherapy; stress; older adults; stress-related change
MeSH Terms: interventions — Odorants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- stress reducing aroma (Experimental): aroma with reported stress reducing effects
  Interventions: Other: aroma
- Placebo aroma 1 (Placebo Comparator)
  Interventions: Other: aroma
- Placebo aroma 2 (Placebo Comparator)
  Interventions: Other: aroma

INTERVENTIONS:
Other: aroma — Comparison of known stress reducing aroma to placebo aromas without stress-reducing effects
  Other Names: lavandula angustifolia; cocos nucifera; aqua destillata

SUMMARY:
The study purpose is to evaluate efficacy of stress-reducing aromatherapy and learn about how aromatherapy works.

DETAILED DESCRIPTION:
The study purpose is to evaluate efficacy of stress-reducing aromatherapy and learn about how aromatherapy works by comparing participants' physiologic responses to laboratory challenge tasks with and without experiencing aromatherapy.

ELIGIBILITY:
Inclusion Criteria:

* in good physical and cognitive health
* reporting moderate level of stress
* able to perceive aromas
* able to understand and follow study instructions

Exclusion Criteria:

* taking medications affecting central nervous system (CNS) function or physiologic measures (e.g. steroids or neuroleptics)
* reporting smell sensitivities or allergies
* smoking presently or in the past less than one year prior to enrollment

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry S Oken, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Chamine I, Oken BS. Aroma Effects on Physiologic and Cognitive Function Following Acute Stress: A Mechanism Investigation. J Altern Complement Med. 2016 Sep;22(9):713-21. doi: 10.1089/acm.2015.0349. Epub 2016 Jun 29. PMID 27355279
- [Result] Chamine I, Oken BS. Expectancy of stress-reducing aromatherapy effect and performance on a stress-sensitive cognitive task. Evid Based Complement Alternat Med. 2015;2015:419812. doi: 10.1155/2015/419812. Epub 2015 Jan 31. PMID 25802539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 212 people potentially interested in the study were evaluated for eligibility between 2010 and 2012. The potential participants were referred by clinicians from the university sleep clinic or learned about the study from the IRB-approved study information posted around the university, or published on social media.
Groups:
- Detectable Placebo Aroma: Coconut: Detectable placebo aroma:organic virgin coconut (Cocos nucifera) base oil (The Ananda Apothecary, Boulder, CO) diluted in 15 ml of grapeseed carrier oil (Now Foods, Bloomingdale, IL) and mixed until solution appeared clear.
  During the visit, three drops of the aroma solution were placed on a 5 x 5 mm cotton pad. The pad was then fixed to a small piece of transparent odor free tape that was attached to the participant's nose so that the pad infused with the aroma came to the midpoint between the participant's nose and upper lip. The cotton pad remained attached until the end of testing portion of the visit, but the aroma was not replenished during the testing.
- Stress Reducing Aroma: Lavender: One drop (using a dropper) of organic lavender (Lavandula angustifolia) essential oil (Mountain Rose Herbs, Eugene, OR) was diluted in 15 ml of grapeseed carrier oil (Now Foods, Bloomingdale, IL).
  During the visit, three drops of the aroma solution were placed on a 5 x 5 mm cotton pad. The pad was then fixed to a small piece of transparent odor free tape that was attached to the participant's nose so that the pad infused with the aroma came to the midpoint between the participant's nose and upper lip. The cotton pad remained attached until the end of testing portion of the visit, but the aroma was not replenished during the testing.
- Undetectable Placebo Aroma: Water: For the undetectable placebo aroma, distilled water was used to provide the appearance of essential oil while emitting no odor and producing no effects typically attributed to aromatherapy.
Period: Overall Study
Arm/Group | Detectable Placebo Aroma: Coconut | Stress Reducing Aroma: Lavender | Undetectable Placebo Aroma: Water
Started | 31 | 31 | 30
Completed | 31 | 31 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Aroma 1: aroma: Comparison of known stress reducing aroma to placebo aromas without stress-reducing effects.
  Coconut aroma with pleasant odor but no reported stress-reducing effects
- Placebo Aroma 2: aroma: Comparison of known stress reducing aroma to placebo aromas without stress-reducing effects.
  Distilled water: substance with no odor or stress-reducing effects
- Total: Total of all reporting groups
Arm/Group | Stress Reducing Aroma | Placebo Aroma 1 | Placebo Aroma 2 | Total
Number analyzed (Participants) | 31 | 31 | 30 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (6.6) | 57.9 (6.0) | 57.3 (5.9) | 58.0 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 23 | 73
  Male | 7 | 5 | 7 | 19
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 31 | 92

OUTCOME MEASURES:

1. Primary Outcome: Percent of Baseline Level of Salivary Cortisol
Description: Percent of baseline level of salivary cortisol (values greater than baseline indicate increased stress)
Time Frame: assessed at baseline (60 min prior to aroma exposure and stress), stress battery (30 min after aroma exposure and during stress), post-stress (60 min after completing stress battery)
Measure: Mean (Standard Error); unit: percentage of baseline cortisol level
Groups:
- Stress Reducing Aroma:Lavender: Lavender aroma with reported stress reducing effects
- Detectable Placebo Aroma: Coconut: Coconut aroma with pleasant detectable smell but without known stress-reducing effects.
- Undetectable Placebo Aroma: Water: Distilled water: substance without smell or known stress-reducing effects
Arm/Group | Stress Reducing Aroma:Lavender | Detectable Placebo Aroma: Coconut | Undetectable Placebo Aroma: Water
Number analyzed (Participants) | 31 | 31 | 30
percentage of baseline cortisol level
  stress battery | 170.8 (31.3) | 224.7 (30.8) | 274.7 (31.9)
  post-stress | 106.4 (70.6) | 187.3 (69.5) | 131.2 (71.9)
Statistical Analysis 1: Comparison: Stress Reducing Aroma:Lavender vs Detectable Placebo Aroma: Coconut vs Undetectable Placebo Aroma: Water; The null hypothesis stated that there were no differences between the groups in cortisol level trajectory over time; Test type: Other; p = .005, ANCOVA — The p value was adjusted for multiple comparisons using false discovery rate; Repeated-measures ANOVA with time (stress, post-stress) as a within factor and aroma (lavender, coconut, water) as a between-group factor was used

2. Secondary Outcome: Electroencephalography (EEG) Frontal Asymmetry
Description: EEG frontal asymmetry (FA) is used to assess emotional state. EEG FA processing was completed by averaging local reference EEG filtered offline from 0.1 to 70 Hz (with 60 Hz notch filter). 5-min data periods during each time were segmented into 2 seconds epochs, and the semi-automatic artifact rejection was applied. The remaining artifact-free epochs were subjected to Fast Fourier Transform (FFT) . The power spectra for individual epochs were averaged, and the measures of EEG spectral density were obtained for alpha band (8 -12.99 Hz). Square root values of power were used, and frontal hemispheric asymmetry was calculated as ((L-R)/(L+R))*100, where L and R are square root values at the homologous left and right hemisphere sites (using local average reference values at F3 and F4). With this calculation, FA negative values reflect lower alpha power (higher activation) in the left hemisphere linked to a more positive mood. This is a unit-free measure.
Time Frame: assessed at baseline (60 min prior to aroma exposure and stress), at the onset of aromatherapy exposure, stress battery (30 min after aroma exposure and during stress), post-stress (60 min after completing stress battery)
Population: All participants had EEG recordings during their visit. However, some EEG data were lost due to electrode malfunction or unusable due to presence of too much noise. The data loss was similar in all study groups.
Measure: Mean (Standard Error); unit: unitless
Groups:
- Stress Reducing Aroma: Lavender: Aroma with reported stress reducing effects
- Detectable Placebo Aroma: Coconut: Coconut: aroma with detectable pleasant smell but without known stress-reducing effects
- Undetectable Placebo Aroma: Water: Distilled water: substance with no smell or known stress-reducing effects.
Arm/Group | Stress Reducing Aroma: Lavender | Detectable Placebo Aroma: Coconut | Undetectable Placebo Aroma: Water
Number analyzed (Participants) | 27 | 27 | 27
unitless
  Baseline | .013 (.027) | .006 (.026) | .036 (.028)
  Aromatherapy exposure onset | .005 (.028) | -.014 (.027) | .064 (.029)
  Stress battery | .031 (.027) | -.001 (.026) | .066 (.029)
  Post-stress | .009 (.026) | .037 (.025) | .089 (.027)

3. Secondary Outcome: Cognitive Performance: Percent Change From Baseline in Digit Span Backward Task Score
Description: Percent change from baseline in cognitive performance score on the Digit Span Backward (DSB) task. DSB scores range from 0 to 16, with greater scores indicative of better cognitive function. Positive change from baseline indicates better functioning.
Time Frame: Baseline (60 min prior to aroma exposure and stress), post-stress (60 min after completing stress battery)
Measure: Mean (Standard Deviation); unit: Percent change from baseline in DSB task
Groups:
- Detectable Placebo Aroma: Coconut: Coconut: aroma with detectable pleasant odor but no reported stress-reducing effects
- Undetectable Placebo Aroma: Water: Distilled water: substance with no odor or known stress-reducing effects.
Arm/Group | Stress Reducing Aroma: Lavender | Detectable Placebo Aroma: Coconut | Undetectable Placebo Aroma: Water
Number analyzed (Participants) | 31 | 31 | 30
Percent change from baseline in DSB task | 15.24 (4.09) | -.37 (4.09) | 0.92 (4.15)
Statistical Analysis 1: Comparison: Stress Reducing Aroma: Lavender vs Detectable Placebo Aroma: Coconut vs Undetectable Placebo Aroma: Water; Test type: Other; p = .01, ANCOVA — P value was adjusted for multiple comparisons using false discovery rate; A 3 (lavender, coconut, water) by 2 ( prime, no prime) Analysis of Covariance (ANCOVA), with years of education as a covariate was used

ADVERSE EVENTS:
Time Frame: The subjects actively participated in the study during one visit, approximately 4 hours in length. The adverse event data were collected for each subject during and immediately after their active study participation. The subjects were encouraged to call if they experienced any adverse events they thought might be related to the study. The overall study period of active enrollment and participation lasted between years 2010 and 2012.
Groups:
- Detectablle Placebo Aroma: Coconut: Aroma with pleasant odor but no known stress-reducing effects
- Undetectalbe Placebo Aroma: Water: Distilled water: substance with no odor or known stress-reducing effects
Arm/Group | Stress Reducing Aroma: Lavender | Detectablle Placebo Aroma: Coconut | Undetectalbe Placebo Aroma: Water
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 1/31 | 0/31 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stress Reducing Aroma: Lavender (N=31) | Detectablle Placebo Aroma: Coconut (N=31) | Undetectalbe Placebo Aroma: Water (N=30)
Headache after study participation (Product Issues) | 1 (1) | 0 (0) | 0 (0) — One participant reported mild headache after study participation that can be related to stress inherent in the study visit or could be due to reacting to aroma. The event resolved on its own after the end of the visit.

LIMITATIONS AND CAVEATS:
Sample included well-educated people over 50 interested in aromatherapy (mostly female). The essential oil and placebo aromas preparations were study-specific.The results are most relevant to the doses and preparations of the aroma stimuli we used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No